CLINICAL TRIAL: NCT05367973
Title: A Phase 1/2,, Open-label, Parallel Group Study to Evaluate the Safety and Pharmacokinetics of DARE-HRT1 (80ug Estradiol/4 mg Progesterone and 160ug Estradiol/8 mg Progesterone Intravaginal Rings) Over 12 Weeks in Healthy Postmenopausal Women
Brief Title: Study of DARE-HRT1 Over 12 Weeks in Healthy PostMenopausal Women
Acronym: DARE-HRT1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DARE-HRT1-002
Record Dates: First submitted 2022-05-02; First posted 2022-05-10 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Vulvovaginal Atrophy; Vasomotor Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVR: Estradiol 80 ug/day + progesterone 4mg/day (Experimental): 12-week IVR 80/4
  Interventions: Device: IVR Dose 1
- IVR Estradiol 160 ug/day + progesterone 8 mg/day (Experimental): 12-week IVR 160/8
  Interventions: Device: IVR Dose 2

INTERVENTIONS:
Device: IVR Dose 1 — Estradiol 80 ug/day + progesterone 4 mg/day
  Arms: IVR: Estradiol 80 ug/day + progesterone 4mg/day
Device: IVR Dose 2 — Estradiol 160 ug/day + progesterone 8 mg/day
  Arms: IVR Estradiol 160 ug/day + progesterone 8 mg/day

SUMMARY:
Randomized, Open-label 2-arm, parallel group study in approximately 20 healthy postmenopausal women to assess the safety of DARE-HRT1 Intravaginal Rings in two different dose strengths and the PK of progesterone and estradiol from the Intravaginal Rings.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women with a body mass index (BMI) ≥ 18 and ≤ 38 kg/m2. BMI = weight (kg)/(height [m])2

   Postmenopausal is defined as 12-months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy (although participants who have had a hysterectomy are not eligible for this study).

   The investigator will need to determine if a participant's BMI falling within the obese-severely obese range could potentially interfere with the protocol-required procedures, specifically the pelvic examinations described in Inclusion Criterion #2. Any participant whose BMI is determined to fall into this category should be excluded from trial participation.
2. Normal cervix, vagina, uterus, and adnexa based on speculum examination and bimanual examination.
3. Normal transvaginal ultrasound, and endometrial biopsy results as follows:

   * If endometrial thickness is ≤ 4.0 mm in a participant without postmenopausal vaginal bleeding, an endometrial biopsy is not indicated for the purposes of screening,
   * If endometrial thickness is > 4.0 mm ≤ 6.0 mm in a participant without postmenopausal vaginal bleeding, an acceptable result from an evaluable screening endometrial biopsy, evaluated by a pathologist, is required for inclusion into the study. Tissue must be read as benign, inactive, or atrophic endometrium by at least 1 pathologist,
4. Current on all Australian screening requirements for cervical cancer.
5. Able and willing to correctly and independently complete all study procedures.
6. Able and willing to stop any ongoing HRT in accordance with the appropriate washout periods (see Section 4.1 for washout requirements). Participants who are using HRT that requires more than 8 weeks to wash out (e.g., progestogen implants or progestogen injectable drug therapy, estrogen alone injectable drug therapy or estrogen pellet therapy) will not be eligible.
7. Able to read, understand, and provide written informed consent after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures.
8. Normal mammogram report within 24 months of screening.

Exclusion Criteria:

1. Prior abnormal cervical screening test or Papanicolaou result within 2 years of screening. Participant can have atypical squamous cells of undetermined significance, if human papillomavirus negative.
2. Participants with any self-reported active sexually transmitted disease and/or evidence of infection based on vaginal visual examination by the investigator.
3. Participants with a urinary tract infection during screening as assessed by urine dipstick test with abnormal test findings (any positive result for leukocytes AND any positive result for nitrites).
4. Have a history of endometrial hyperplasia or cervical or uterine carcinoma.
5. Participants with indwelling catheters or requiring intermittent catheterization.
6. Participants with multiple or unsuccessful (e.g., still having symptoms) pelvic reconstructive surgery, or who suffer from pelvic relaxation.
7. Participants who have had a hysterectomy.
8. Participants taking any estrogen and/or progesterone products who are not willing to stop this treatment during their participation in this trial (see Section 4.1 for washout requirements). Participants who are using HRT that requires more than 8 weeks to wash out (e.g., progestogen implants or progestogen injectable drug therapy, estrogen alone injectable drug therapy or estrogen pellet therapy) will not be eligible.
9. Participants with concomitant use of personal lubricants (water-based lubricants are allowed) or any intravaginal product or medication, either by prescription or over-the-counter (OTC) (e.g., Femring [estradiol acetate vaginal ring], ESTRING® [estradiol vaginal ring]) with the exception of those who agree not to use these products during the IVR use period.
10. Self-reported or observed vaginal irritation unrelated to VVA; vaginal, vulvar, or cervical lesions, undiagnosed vaginal bleeding; or tenderness.
11. Participants with a finding of clinically significant uterine fibroids at screening.
12. Participants with a known hypersensitivity to progesterone, estradiol, Femring, or the components of the IVR (e.g., ethylene vinyl acetate).
13. Participants with prior pelvic malignancies.
14. Participants with a history of any severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or study treatment administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the participant inappropriate for entry into the trial. This includes but is not limited to the following:

    1. Human immunodeficiency virus (HIV) infection (confirmed by medical history/ serology testing),
    2. Active chronic hepatitis B or hepatitis C infection including hepatitis B surface antigen and hepatitis C antibody positive participants with or without abnormal liver enzymes (confirmed by medical history/serology testing),
    3. Concurrent neurodegenerative disease,
    4. Cardiovascular: uncontrolled hypertension, unstable angina, myocardial infarction or symptomatic congestive heart failure within the past 6 months, serious uncontrolled cardiac arrhythmia, use of Class 1 antiarrhythmic medications, or history of venous thromboembolism or stroke,
    5. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of the protocol,
    6. Participants with known thrombophilias may not participate in this study because estrogen-based products are contraindicated for them,
    7. Symptomatic bacterial vaginosis.
15. Fasting triglyceride of > 3.39 mmol/L and/or total cholesterol of > 7.77 mmol/L.
16. Aspartate aminotransferase or alanine aminotransferase > 1.5 times the upper limit of normal.
17. Fasting glucose > 6.94 mmol/L.
18. Evidence of current alcohol or drug abuse in the past 60 days including a positive result from the urine drugs of abuse or alcohol screen, or history of drug or alcohol dependence in the last 2 years, as assessed by principal investigator. Alcohol abuse is defined as greater than 14 standard units/week for females and drug abuse is defined as known psychiatric or substance abuse disorder that would interfere with participation with the requirements of this study, including current use of any illicit drugs. Use of medical cannabis is not exclusionary.
19. Participation in any other investigational drug or device trial in which administration of an investigational study drug/device occurred within 30 days or placement of a non-drug eluting medical device within 15 days prior to screening.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - PARC Clinical Research, Adelaide, Southern Australia
  - Keogh Institute for Medical Research, Nedlands, Western Australia

REFERENCES:
- [Derived] Thurman A, Hull ML, Stuckey B, Hatheway J, Zack N, Mauck C, Friend D. A phase 1/2, open-label, parallel group study to evaluate the preliminary efficacy and usability DARE-HRT1 (80 mug estradiol/4 mg progesterone and 160 mug estradiol/8 mg progesterone intravaginal RinGSM) over 12 weeks in healthy postmenopausal women. Menopause. 2023 Sep 1;30(9):940-946. doi: 10.1097/GME.0000000000002230. Epub 2023 Aug 7. PMID 37625088
- [Derived] Thurman A, Hull ML, Stuckey B, Hatheway J, Zack N, Mauck C, Friend D. A phase 1/2, open-label, parallel group study to evaluate the safety and pharmacokinetics of DARE-HRT1 (80 mug estradiol/4 mg progesterone and 160 mug estradiol/8 mg progesterone intravaginal rings) over 12 weeks in healthy postmenopausal women. Menopause. 2023 Aug 1;30(8):817-823. doi: 10.1097/GME.0000000000002210. Epub 2023 Jun 20. PMID 37339390

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day
Started | 11 | 10
Completed | 11 | 8
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (3.41) | 59.0 (4.74) | 58.8 (4.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 11 | 10 | 21
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (3.53) | 28.9 (4.62) | 27.3 (4.26)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: To assess the safety and tolerability of DARE-HRT1 Intravaginal rings
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day
Number analyzed (Participants) | 11 | 10
Participants | 11 | 10

2. Primary Outcome: Determination of Maximum Plasma Concentration of Progesterone (Cmax) Per Cycle
Description: To describe the Pharmacokinetic parameters of dose combinations (Estradiol 80 ug/progesterone 4/mg day and Estradiol 160 ug/progesterone 8/mg day)
Time Frame: 12 weeks (3- 28 day cycles)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 1; IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 2; IVR: Estradiol 80 ug/Day + Progesterone 4 mg/Day Cycle 3: 28 day IVR 80/4
  IVR Dose 1: Estradiol 80 ug/day + progesterone 4 mg/day
- IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day Cycle 1; IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 2; IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 3: 28 day IVR 160/8
  IVR Dose 2: Estradiol 160 ug/day + progesterone 8 mg/day
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 1 | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 2 | IVR: Estradiol 80 ug/Day + Progesterone 4 mg/Day Cycle 3 | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day Cycle 1 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 2 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 3
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 8
ng/mL | 5.16 (43.83) | 2.40 (36.8) | 2.71 (30.95) | 8.45 (37.75) | 3.46 (15.73) | 3.38 (10.01)

3. Primary Outcome: Determination of Time That Maximum Progesterone Plasma Concentration Was Observed (Tmax)
Description: as for outcome 2
Time Frame: 12 weeks (3- 28 day cycles)
Measure: Median (Full Range); unit: hours
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 1 | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 2 | IVR: Estradiol 80 ug/Day + Progesterone 4 mg/Day Cycle 3 | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day Cycle 1 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 2 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 3
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 8
hours | 23.23 [7.85 to 24.20] | 24.08 [0.50 to 48.30] | 0.500 [.050 to 23.03] | 23.25 [23.00 to 24.82] | 23.67 [1.00 to 47.95] | 4.00 [0.48 to 48.17]

4. Primary Outcome: Determination of Progesterone Steady-state Concentration (Css) Per Cycle
Description: as for outcome 2
Time Frame: 12 weeks (3- 28day cycles)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 1 | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 2 | IVR: Estradiol 80 ug/Day + Progesterone 4 mg/Day Cycle 3 | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day Cycle 1 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 2 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 3
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 8 | 7
ng/mL | 1.06 (25.57) | 1.08 (27.49) | 1.21 (26.72) | 1.83 (26.10) | 1.68 (13.39) | 1.78 (15.41)

5. Other Pre Specified Outcome: Evaluation of Responses to The Menopause-Specific Quality-of-Life Questionnaire (MENQOL)
Description: To assess usability and participant tolerability of the DARE-HRT1 Intravaginal Ring comparing total questionnaire score from baseline to end of study with a decrease in score showing improvement.
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Evaluation of Vaginal Cytology
Description: To conduct a preliminary evaluation of the effect of the DARE-HRT1 intravaginal ring on Vulvarvaginal atrophy
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Evaluation of Vaginal pH
Description: To conduct a preliminary evaluation of the effect of the DARE-HRT1 intravaginal ring on Vulvarvaginal atrophy
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Evaluation of Most Bothersome Symptom Via Subject Self Report
Description: To conduct a preliminary evaluation of the effect of the DARE-HRT1 intravaginal ring on Vasomotor Symptoms (VMS)
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Primary Outcome: Determination of Time That Maximum Estradiol Plasma Concentration Was Observed (Tmax)
Description: as for outcome 2
Time Frame: 12 weeks (3- 28 day cycles)
Measure: Median (Full Range); unit: hours
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 1 | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 2 | IVR: Estradiol 80 ug/Day + Progesterone 4 mg/Day Cycle 3 | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day Cycle 1 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 2 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 3
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 8
hours | 24.20 [22.07 to 48.05] | 47.48 [23.28 to 167.08] | 47.26 [23.03 to 48.43] | 47.09 [23.07 to 48.85] | 47.95 [23.23 to 170.87] | 47.26 [23.07 to 48.23]

10. Primary Outcome: Determination of Maximum Plasma Concentration of Estradiol (Cmax) Per Cycle
Description: as for outcome 2
Time Frame: 12 weeks (3- 28 day cycles)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 1 | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 2 | IVR: Estradiol 80 ug/Day + Progesterone 4 mg/Day Cycle 3 | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day Cycle 1 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 2 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 3
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 8
pg/mL | 68.29 (27.29) | 41.67 (35.91) | 44.56 (21.00) | 107.76 (34.17) | 66.89 (31.66) | 71.06 (34.48)

11. Primary Outcome: Determination of Estradiol Steady-state Concentration (Css) Per Cycle
Description: as for outcome 2
Time Frame: 12 weeks (3- 28day cycles)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 1 | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day Cycle 2 | IVR: Estradiol 80 ug/Day + Progesterone 4 mg/Day Cycle 3 | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day Cycle 1 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 2 | IVR: Estradiol 160 ug/Day + Progesterone 8mg/Day Cycle 3
Number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 8
pg/mL | 21.87 (36.92) | 22.55 (22.83) | 21.79 (20.15) | 37.28 (22.17) | 36.43 (24.00) | 37.52 (27.68)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day (N=11) | IVR Estradiol 160 ug/Day + Progesterone 8 mg/Day (N=10)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2) | 4 (6)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Postmenopausal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 2 (4)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (9) | 5 (11)
Sensory distrubance (Nervous system disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 2 (6) | 2 (5)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI are not allowed to publish without prior approval from Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT05367973/Prot_SAP_000.pdf